CLINICAL TRIAL: NCT06264596
Title: The Effect of Epinephrine in Irrigation Fluid for Visualization During Ankle Arthroscopy: A Randomized Blinded Controlled Trial
Brief Title: Epinephrine in Irrigation Fluid for Visualization During Ankle Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never started. PI is leaving institution.
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2310-72
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Intraoperative Bleeding
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Concealed irrigation bags
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epinephrine (Experimental): The epinephrine group will have two 3-L normal saline solution bags prepared for each case with 1 mL of 1:1000 epinephrine in each bag (epinephrine concentration 1:3,000,000 for each bag).
  Interventions: Drug: Epinephrine; Procedure: Normal Saline irrigation fluid
- Normal saline (Placebo Comparator): The control group will have two 3-L normal saline solution bags prepared with no additive
  Interventions: Procedure: Normal Saline irrigation fluid

INTERVENTIONS:
Drug: Epinephrine — The epinephrine group will have two 3-L normal saline solution bags prepared for each case with 1 mL of 1:1000 epinephrine in each bag
  Other Names: Epinephrine in irrigation fluid
  Arms: Epinephrine
Procedure: Normal Saline irrigation fluid — The control group will have two 3-L normal saline solution bags prepared with no additive

SUMMARY:
The purpose of this study is to evaluate the effect of epinephrine in irrigation fluid for visual clarity in ankle arthroscopic surgery.

DETAILED DESCRIPTION:
The primary outcomes are:

* visual clarity during ankle arthroscopic surgery, which will be evaluated by visual analog scale from 0-10,
* and the intraoperative surgeon's discomfort related to bleeding, that will be measured by visual numeric rating scale from 0-3.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females ages over 18 years
* Patients who undergo ankle arthroscopic surgery
* Patients who are able to read and give informed consent on their own behalf

Exclusion Criteria:

* Patients with any known cardiac diseases
* Uncontrolled hypertension (> 180/110 mmHg)
* Revision case
* Younger than 18 years of age
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
visual clarity during ankle arthroscopic surgery, which will be evaluated by visual analog scale | intraoperative
  visual analog scale from 0-10
surgeon's discomfort related to bleeding, measured by visual numeric rating scale | intraoperative
  visual numeric rating scale 0-3

CONTACTS AND LOCATIONS:
Overall Officials: Wonyong Lee, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No